CLINICAL TRIAL: NCT04276428
Title: A Multiple-Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY3209590 in Japanese Patients With Type 2 Diabetes Mellitus
Brief Title: A Study of LY3209590 in Japanese Participants With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 16983; I8H-JE-BDCK (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-02-18; First posted 2020-02-19 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin degludec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- LY3209590 (Experimental): LY3209590 administered subcutaneously (SC).
  Interventions: Drug: LY3209590
- Insulin Degludec (Active Comparator): Insulin degludec administered SC.
  Interventions: Drug: Insulin Degludec

INTERVENTIONS:
Drug: LY3209590 — Administered SC.
  Arms: LY3209590
Drug: Insulin Degludec — Administered SC.
  Arms: Insulin Degludec

SUMMARY:
The main purpose of this study is to evaluate the safety of a study drug known as LY3209590 in Japanese participants with type 2 diabetes. Side effects and tolerability will be documented. Blood samples will be taken to compare how the body handles the drug and how it affects blood sugar levels. The study will last almost five months for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Have type 2 diabetes mellitus (T2DM) for at least 1 year
* Have received a stable daily dose of basal insulin at screening
* Have hemoglobin A1c (HbA1c) greater than or equal to (≥)6.5 percent (%) and less than or equal to (≤)10.0% at screening
* Have a body mass index greater than (>)18.5 and ≤40.0 kilograms per square meter (kg/m²) at screening

Exclusion Criteria:

* Have received a total daily dose of insulin >1.2 units per kilogram (U/kg) of body weight at screening
* Have received insulins except for basal insulins
* Have received sulfonylurea at more than half of the maximum approved dose level
* Have a history of multiple and/or severe allergies to drugs or foods or a history of severe anaphylactic reaction or history of significant atopy
* Have had more than 1 episode of severe hypoglycemia within 6 months before entry

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2020-11-28 (Actual); Study Completion 2020-11-28 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline through Day 85
  A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Drug-Plasma-Concentration-Versus-Time Curve from Time Zero to 168 Hours Postdose (AUC[0-168]) of LY3209590 | Predose on Day 1 through Day 85
  PK: AUC(0-168) of LY3209590
Pharmacodynamics (PD): Change from Baseline in Fasting Plasma Glucose | Day 1 through Day 85
  PD: Change from Baseline in Fasting Plasma Glucose

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- Japan (3):
  - Clinical Research Hospital Tokyo, Shinjuku-ku, Jp-13
  - P-one clinic, Hachiōji, Tokyo
  - Yokohama Minoru Clinic, Yokohama

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nasu R, Oura T, Ohwaki K, Imori M, Furihata K. Pharmacokinetic and Pharmacodynamic Properties of Once-Weekly Insulin Efsitora Alfa in Japanese Patients with Type 2 Diabetes. Diabetes Ther. 2025 Mar;16(3):513-526. doi: 10.1007/s13300-025-01695-x. Epub 2025 Feb 10. PMID 39928225